CLINICAL TRIAL: NCT04040270
Title: 3Hs Family Drama Project
Brief Title: Family Drama Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Boys' and Girls' Clubs Association of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 12-409
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Family Health, Happiness and Harmony; Physical Health
Keywords: Family well-being; Healthy Eating; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Live drama+DVD+Worksheets (Experimental): Primary school students watched an interactive live drama in schools. DVD and worksheets were also distributed to students and asked them to watch the DVD and finish the worksheets with their parents.
  Interventions: Behavioral: Live drama+DVD+Worksheets
- DVD+Worksheets (Experimental): Primary school students were given DVD and worksheets and they were asked to watch the DVD and finish the worksheets with their parents. After the study finished, the students watched the live drama.
  Interventions: Behavioral: DVD+Worksheets
- Waitlist control (No Intervention): Primary school students received no intervention during the 4-week study period. After the study finished, the students watched the live drama, and DVD with worksheets were distributed to students and they were encouraged to share with their parents.

INTERVENTIONS:
Behavioral: Live drama+DVD+Worksheets — Interactive live drama was proposed to enhance memories of the audience of health promotion programmes.
  The interactive live drama and DVD conveyed educational information on healthy living habits (including physical activity and healthy eating) as well as the importance and suggested methods to enhance family well-being. Students were encouraged to share the information on healthy living habits and watched the DVD with their parents.
  Worksheets were given to all students and encouraged to finish the worksheets with their parents.
  Arms: Live drama+DVD+Worksheets
Behavioral: DVD+Worksheets — The DVD conveyed educational information on healthy living habits (including physical activity and healthy eating) as well as the importance and suggested methods to enhance family well-being. Students were encouraged to share the information on healthy living habits and watched the DVD with their parents.
  Worksheets were given to all students and encouraged to finish the worksheets with their parents.
  Arms: DVD+Worksheets

SUMMARY:
A harmonious family relationship has significant effects on the psychological well-being and development of children. Good communication between parents and children is a crucial element for family health, happiness and harmony. However, communication within Hong Kong families is vastly inadequate partly due to our busy urban lifestyle.

The 3Hs Family Drama Project I was to promote health, happiness, harmony (3Hs), healthy eating and physical activity in primary school students. Students watched interactive live drama in schools and were given DVD and worksheets. Students were encouraged to watch the DVD with other family members at home. This study was to evaluate the effectiveness of interactive live drama, DVD and worksheet.

DETAILED DESCRIPTION:
3Hs Family Drama Project was an intervention to enhance the 3Hs through increasing interaction and communication between parents and children. Healthy eating and physical activity were also promoted. The drama project staged 100 drama performances in primary schools during the 2012-13 school year. The main targets were Primary 4 to 6 (P4-6) students and their families. Group A students would watch the live drama in school and were encouraged to watch the DVD and finish worksheets with their parents, while group B students would be given a DVD and worksheets and were encouraged to watch the DVD and finish the worksheets with their parents.

The goals of the study were to evaluate the effectiveness of the project to enhance health, happiness, harmony (3Hs), healthy eating and physical activity and participants' satisfaction levels towards the drama project.

Quantitative assessments were used to evaluate the effectiveness and the satisfaction of the project. Questionnaire was distributed to assess the immediate and short-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Primary 4 to 6 students in participating primary schools.

Exclusion Criteria:

* Students who cannot read Chinese.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7453 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Change in family health, happiness and harmony (3Hs) | baseline and 4 weeks
  Health, happiness and harmony (3Hs) were assessed by family well-being scale. Perceived family harmony and health were measured by 2 questions on a scale ranging from 1 to 5, whereas perceived family happiness was measured by a single question on a scale ranging from 1 to 4. The higher score the better.

SECONDARY OUTCOMES:
Change in parent-child interactions | baseline, 1 week and 4 weeks
  Students were asked whether they performed the 12 mentioned activities (e.g. watching movies with parents) in the past 7 days.
Change in fruit and vegetable consumption | baseline, 1 week and 4 weeks
  Students were asked to report the number of days (0-7) of consuming at least 2 servings of fruit and 3 servings of vegetables in the past 7 days.
Change in behavior on moderate-to-vigorous physical activity | baseline, 1 week and 4 weeks
  Students were asked to report the number of days (0-7) of at least 60 minutes moderate-to-vigorous physical activity in the past 7 days.
Satisfaction towards the live drama and take-home DVD | 1 week and 4 weeks
  Students were asked to rate the live drama, DVD on a scale ranging from 1 to 5. The higher score the more satisfied.
Change in family health, happiness and harmony (3Hs) | baseline and 1 week
  Health, happiness and harmony (3Hs) were assessed by family well-being scale. Perceived family harmony and health were measured by 2 questions on a scale ranging from 1 to 5, whereas perceived family happiness was measured by a single question on a scale ranging from 1 to 4. The higher score the better.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Yin Ho, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Local primary schools, Hong Kong, Hong Kong